CLINICAL TRIAL: NCT03329560
Title: Safety of Fecal Microbiota Transplant Using Oral Encapsulated PRIM-DJ2727 in HIV-infected Persons on Antiretroviral Therapy
Brief Title: Safety of FMT Using Oral Encapsulated PRIM-DJ2727 in HIV
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Netanya Utay, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-17-0782
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Oral fecal microbiota transplantation (Experimental): All subjects will receive one dose per week for 6 weeks (6 total doses) of PRIM-DJ2727 oral capsules containing lyophilized microbiota product derived from 150 grams of healthy donor stool.
  Interventions: Biological: Oral fecal microbiota transplantation

INTERVENTIONS:
Biological: Oral fecal microbiota transplantation — All subjects will receive one dose per week for 6 weeks (6 total doses) of PRIM-DJ2727 oral capsules containing lyophilized microbiota product derived from 150 grams of healthy donor stool.
  Other Names: PRIM-DJ2727

SUMMARY:
The purpose of this study is to determine whether oral fecal microbiota transplantation (FMT) is safe for people with human immunodeficiency virus (HIV) infection.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, documented by any licensed HIV test
* Male subjects ≥ 18 years of age
* Identify as MSM (men who have sex with men)
* Currently on continuous ART for ≥24 weeks prior to study entry with no change in the ART regimen within the 12 weeks prior to study
* Ability and willingness of the participating subject to sign the informed consent form
* No plan to change ART regimen for the study duration
* Screening CD4+ cell count >350 cells/mm3 obtained within 45 days prior to study entry
* HIV RNA < 20 copies/ml for ≥12 weeks (1 blip of < 500 copies/ml will be permitted)
* Absolute neutrophil count ≥ 1000 cells/mm3

Exclusion Criteria:

* Initiation of ART during acute/early HIV infection (within 6 months of HIV seroconversion)
* Co-infection with Hepatitis B (positive HBsAg or positive HBcAb total with detectable HBV DNA levels) or Hepatitis C (positive HCV IgG with detectable HCV RNA levels)
* Use of antibiotics 60 days prior to the study entry
* Use of investigational therapies or vaccines 60 days prior to the study entry
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to entry
* Cirrhosis, inflammatory bowel disease, total colectomy, colon or rectal anastomosis, bowel resection, or current colostomy
* Diabetes mellitus
* Any episode of acute or persistent diarrhea within 60 days prior to study entry
* Use of any of the following medications/products for more than 3 consecutive days within the 60 days prior to study entry: Immunosuppressives, Immune modulators, Antineoplastic agents (except for topical agents for skin cancer), Probiotics and prebiotics (supplements and products).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events related to study drug | 52 weeks
Cumulative of adverse events related to study drug | 52 weeks
Severity of adverse events related to study drug | 52 weeks
  Severity of adverse events will be based on Division of AIDS (DAIDS) grading criteria.

SECONDARY OUTCOMES:
Change in the intestinal microbiome diversity | week 0, week 6
Change in the intestinal microbiome abundance of genera | week 0, week 6
Change in systemic inflammation as assessed by interleukin 6 (IL-6) levels | week 0, week 6
Change in microbial translocation as assessed by soluble cluster of differentiation (CD14) levels | week 0, week 6
Change in gut barrier integrity as assessed by intestinal fatty acid binding protein (I-FABP) | week 0, week 6

CONTACTS AND LOCATIONS:
Overall Officials: Netanya S Utay, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Thomas Street Health Center, Houston, Texas, United States

REFERENCES:
- [Derived] Utay NS, Monczor AN, Somasunderam A, Lupo S, Jiang ZD, Alexander AS, Finkelman M, Vigil KJ, Lake JE, Hanson B, DuPont HL, Arduino RC. Evaluation of Six Weekly Oral Fecal Microbiota Transplants in People with HIV. Pathog Immun. 2020 Dec 30;5(1):364-381. doi: 10.20411/pai.v5i1.388. eCollection 2020. PMID 33501400